CLINICAL TRIAL: NCT01475747
Title: Systolic Pressure Intervention Trial (SPRINT)-Factors Affecting Factors Affecting Atherosclerosis Study (FAST)
Brief Title: Systolic Pressure Intervention Trial Factors Affecting Factors Affecting Atherosclerosis Study
Acronym: SPRINTFAST
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Srinvasan Beddhu, MD, Assiociate Professor of Medicine, University of Utah
Other Study IDs: IRB_00049314; R01DK091437-01 (NIH)
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Hypertension; Chronic Kidney Disease
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, plasma and serum samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational - SPRINT trial subjects: Subjects in the Systolic Pressure Intervention Trial (SPRINT) observed to examine factors that affect atherosclerosis in chronic kidney disease

SUMMARY:
Systolic Pressure Intervention Trial (SPRINT) is a large scale randomized trial of ~ 9250 adults aged 50 years or older with high cardiovascular risk sponsored by NIH. The study is designed to recruit 45% of the study population with Chronic Kidney Disease (CKD). The trial will test the effects of low systolic blood pressure (SBP) goal of < 120 mm Hg versus the standard goal of < 140 mm Hg on the primary composite of cardiovascular events and death. One of the pre-specified secondary outcome is the progression of kidney disease. In this ancillary named SPRINT - Factors affecting Atherosclerosis STudy (FAST), the investigators plan to take advantage of the unique opportunities afforded by the parent study to examine issues that are of significant public health importance.

This is an observational study in SPRINT participants. This study will examine mechanistically, the factors affecting the progression of atherosclerosis in CKD.

ELIGIBILITY:
Inclusion Criteria

* Systolic Pressure Intervention Trial (SPRINT) participants

Exclusion Criteria

* Contraindications to MRI (such as intracranial metal prostheses, weight > 300 pounds, claustrophobia and certain types of hardware used in pacemakers, prostheses, etc.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical characteristics of the SPRINT-FAST population will reflect those of the parent study. In this ancillary study, one non-CKD participant (control) will be recruited for each CKD participant (case). SPRINT CKD stratum will likely comprise of those with eGFR between 20-59 ml/min/1.73 m2.
Sampling Method: Non-Probability Sample
Enrollment: 595 (Actual)
Dates: Start 2011-09; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Development Rate of Atherosclerosis | Baseline and 30 months
  Correlation of the presence of CKD and rate of progression of atherosclerosis as assessed by magnetic resonance imaging (MRI) of the carotid artery.

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Beddhu, MD, Principal Investigator — University of Utah
Locations (12):
- United States (12):
  - Stanford University, Palo Alto, California
  - University of Colorado Denver, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Minnesota, Minneapolis, Minnesota
  - Wake Forest University, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Pittsburgh, Pennsylvania
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Beddhu S, Boucher RE, Sun J, Balu N, Chonchol M, Navaneethan S, Chertow GM, Townsend R, Haley W, Cheung AK, Conroy MB, Raj DS, Xu D, George T, Yunis R, Wei G, Canton G, Bates J, Chen J, Papademetriou V, Punzi H, Wiggers A, Wright JT, Greene T, Yuan C. Chronic kidney disease, atherosclerotic plaque characteristics on carotid magnetic resonance imaging, and cardiovascular outcomes. BMC Nephrol. 2021 Feb 24;22(1):69. doi: 10.1186/s12882-021-02260-x. PMID 33627066